CLINICAL TRIAL: NCT01279148
Title: Electromagnetic Tracking of Devices During Interventional Procedures
Status: Withdrawn | Type: Observational
Sponsor: Philips Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: 2010 MCT V7
Record Dates: First submitted 2011-01-10; First posted 2011-01-19 (Estimated); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Biopsy or Ablation Procedures
Keywords: biopsy guidance; tracking device

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Liver Biopsy analyzed as per standard of care
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Biopsy/Ablation - CONTROL GROUP: The tracking device will be placed on the patient's skin at the desired point of entry. Without displaying the PercuNav screen to the physician, a screen capture will be taken to record the approach path. At the point of insertion, the time stamp will be recorded and the start button will be pressed. Once the physician states they are at the defined target a screen capture will be taken on the PercuNav and the distance to target and time stamp will be recorded by pushing the start button again.
- Biopsy/Ablation - STUDY GROUP:: The tracking device will be placed on the patient's skin at the desired point of entry. Without displaying the PercuNav screen to the physician, a screen capture will be taken to record the approach path. The physician will then be un-blinded and shown the PercuNav screen and will correct the desired approach path and another screen capture will be taken. At the point of insertion, the time stamp will be recorded and the start button will be pressed. Once the physician states they are at the defined target a screen capture will be taken on the PercuNav and the distance to target and time stamp will be recorded. At the end of the procedure, and if clinically indicated, a verification "CT" computed tomography scan will be taken with the needle in place and, sent to the PercuNav. Radiation dosage, due to CT imaging, will also be recorded.

SUMMARY:
This prospective, randomized, controlled, parallel-design trial will compare the use of electromagnetic tracking and image guidance during biopsy/ablation procedures verses the typical standard or conventional image guided procedure alone (control). "US" ultrasound-guided biopsies/ablations with or without "CT" computed tomography- imaging will be used to complete the procedures in either the CT suite or a procedure room, at the discretion of the physician, and according to normal local practice patterns.

DETAILED DESCRIPTION:
The study will consist of approximately 300 patients from 1 sites. Each site will have a study group, where the physician will use the electromagnetic tracking system along with "US" ultrasound or "CT" computed tomography to complete the procedure and a control group, where the electromagnetic tracking system will be used, but the physician will be blinded to it and use only the typical, standard, conventional protocol, using US or CT, to complete the procedure. The expected completion time for enrollment is 12 months, but will depend on the ability of each Clinic to enroll patients.

Data and observations will be collected at a total of 2 scheduled appointments (screening and 1 study visit) or based on the current hospital workflow, which may combine these into one patient encounter.

ELIGIBILITY:
Inclusion Criteria:

* Has had a pre-operative CT scan performed and will be undergoing a biopsy or ablation procedure of the chest, abdomen and/or pelvis;
* Is over the age of 18;
* Has the ability to understand and the willingness to sign a written informed consent form, and complies with the protocol;
* Has the ability to follow procedural instructions, including, but not limited to, holding their breath and remaining reasonably motionless during the procedure.

Exclusion Criteria:

* Was precluded from a biopsy/ablation procedure based on standard exclusions;
* Has an adhesive allergy (due to the application of active fiducials with adhesive backing);
* Has a pacemaker or automatic implantable cardiac defibrillator;
* Has a gross body weight above the procedural table limit (typically > 170 kg);
* Is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitals and Out-patient Clinics
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-04; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Target Registration Error | Day 1
  "TRE" Target Registration Error (distance between "virtual" needle position (tracking data) and the actual needle position ("CT" Computed Tomography confirmation scan))

SECONDARY OUTCOMES:
Success of ablation as determined by imaging | 3 months
  Primary effectiveness (success of ablation in local tumor control or success of biopsy in diagnostic biopsy sample). Successful ablation equals complete tumor ablation with a 5mm-1cm margin of normal tissue (if possible; quantified by the lack of enhancement of intravenous contrast material at 3 month follow up CT).

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States